CLINICAL TRIAL: NCT02889315
Title: Assessment of Safety and Efficacy of Implantable Pump (LenusPro) in Patients With Pulmonary Arterial Hypertension Treated With Treprostinil.
Brief Title: LenusPro Pump in PAH Treated With Treprostinil
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Department of Pulmonary Circulation and Thromboembolic Diseases, Medical Center for Postgraduate Med (Other)
Responsible Party: Principal Investigator, Marcin Kurzyna, Marcin Kurzyna, MD, PhD, Department of Pulmonary Circulation and Thromboembolic Diseases, Medical Center for Postgraduate Med
Other Study IDs: 001
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH; treprostinil; LenusPro; implantable device; quality of life
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subcutaneous treprostinil is used to treat pulmonary arterial hypertension (PAH). Due to local pain it causes a deterioration of quality of life or even abandonment of treatment. The aim of this study was to evaluate the safety and quality of life (QoL) in patients treated with treprostinil administration using an implantable Lenus Pro® pump. This is a observational study involving patients with PAH treated with a subcutaneous infusion of treprostinil with intolerable pain at the infusion site, who were therefore referred for pump implantation. Clinical evaluation, including QoL assessment with SF-36 questionnaire was performed at the time of initiating therapy with treprostinil, before and 2-9 months after implantation.

DETAILED DESCRIPTION:
Treprostinil is a prostacyclin analogue, a drug that is widely used to treat pulmonary arterial hypertension (PAH). Its efficacy was confirmed in studies that compared it to placebo and to epoprostenol. Due to stability of treprostinil sodium solution and its relatively long (when compared to prostacyclin) half-life, the drug enabled PAH patients to receive safe long-term treatment. It is administered as a continuous subcutaneous infusion using an insulin pump. In the case of this route of administration, its half-life is about 3 hours. Unfortunately, due to reaction at the infusion site many patients report significant deterioration of quality of life, and some of them (about 5-10%) even abandon treatment . There are trials in progress to find a more convenient method of administration for this drug. The efficacy of oral administration has been uncertain - reports are contradictory, while inhalations remain a valid alternative for patients in a less advanced stage of the disease. Therefore, for patients whose illness is more severe, only continuous parenteral administration of the drug remains an option.

The Lenus Pro® implantable pump appears to be a promising alternative to an external pump. By means of this method, treprostinil sodium is administered as a continuous intravenous infusion, and the drug reservoir is refilled every 28 days. Thermal stability of treprostinil at body temperature was confirmed during a 60-day observation; concentrations of the drug administered intravenously are comparable to subcutaneous administration, and the only differing parameter is a shorter half-life of less than 1 hour. The first experiences with implantable pumps originate in Austria and Germany and present this method of treatment as a milestone in PAH therapy. In Poland, the first implantation of a Lenus Pro® pump took place in 2013 (18).

The aim of this study is an analysis of efficacy and safety of treatment with intravenous treprostinil administered by means of the Lenus Pro® implantable pump.

Prior to pump implantation the subcutaneous dose of treprostinil is escalated up to the highest dose tolerated by a particular patient. The procedure of pump implantation is carried out under general anaesthesia Clinical and haemodynamic evaluation is performed at the time of initiating PAH therapy with treprostinil. Right before and during 2-9 months after Lenus Pro® pump implantation, non-invasive clinical evaluation was made, including: WHO functional class, 6-minute walking test (6MWT), and concentration of NT-proBNP. Additionally patients fill in the SF36 quality of life questionnaire before implantation and 2-9 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Pulmonary Arterial Hypertnesion according to ESC/ERS Guidelines
* treatment with sc treprostinil at stable dose
* poor local tolerance of sc infusion

Exclusion Criteria:

* life expectancy < 6 months
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary arterial hypertension treated with treprostinil in subcutaneous infusion with severe local side effects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2021-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety of transition from subcutaneous delivery do intravenous delivery through LenusPro pump | from implantation to 6 months thereafter
Improvement of QoL caused by changing therapy measured with SF-36 form | from implantation to 6 months thereafter

CONTACTS AND LOCATIONS:
Locations (1):
- European Health Center Otwock, Otwock, Poland

IPD SHARING:
Plan to Share IPD: Undecided